CLINICAL TRIAL: NCT01657799
Title: A Randomized, Double-Blind, Phase 2, Dose-Ranging Study to Evaluate the Safety and Efficacy of Veliparib and Whole Brain Radiation Therapy Versus Placebo and Whole Brain Radiation Therapy in Subjects With Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: Comparison of Veliparib and Whole Brain Radiation Therapy (WBRT) Versus Placebo and WBRT in Adults With Brain Metastases From Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-897; 2011-003618-18 (EudraCT Number)
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-01

CONDITIONS: Brain Metastases From Non-small Cell Lung Cancer
MeSH Terms: interventions — veliparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Veliparib 200 mg BID + WBRT (Experimental): Participants received veliparib 200 mg twice a day (BID) orally concomitantly with whole brain radiation therapy (WBRT). Participants received a total of 30.0 Gy of WBRT given in 10 daily fractions of 3.0 Gy, excluding weekends and holidays.
  Interventions: Drug: Veliparib; Radiation: Whole brain radiation therapy
- Veliparib 50 mg BID + WBRT (Experimental): Participants received veliparib 50 mg twice a day (BID) orally concomitantly with whole brain radiation therapy (WBRT). Participants received a total of 30.0 Gy of WBRT given in 10 daily fractions of 3.0 Gy, excluding weekends and holidays.
  Interventions: Drug: Veliparib; Radiation: Whole brain radiation therapy
- Placebo BID + WBRT (Placebo Comparator): Participants received placebo twice a day (BID) orally concomitantly with whole brain radiation therapy (WBRT). Participants received a total of 30.0 Gy of WBRT given in 10 daily fractions of 3.0 Gy, excluding weekends and holidays.
  Interventions: Drug: Placebo; Radiation: Whole brain radiation therapy

INTERVENTIONS:
Drug: Veliparib — Veliparib capsules for oral administration
  Other Names: ABT-888
  Arms: Veliparib 200 mg BID + WBRT; Veliparib 50 mg BID + WBRT
Drug: Placebo — Placebo to veliparib capsules for oral administration
  Arms: Placebo BID + WBRT
Radiation: Whole brain radiation therapy — 30.0 grays (Gy) of WBRT given in 10 daily fractions of 3.0 Gy each, excluding weekends and holidays

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of veliparib and whole brain radiation therapy in adults with brain metastases from non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Subject must have cytologically or histologically confirmed non-small cell lung cancer
* Subject must have brain metastases demonstrated on a magnetic resonance imaging (MRI) brain scan.
* Subject must be eligible for treatment with WBRT
* Subject must have had adequate hematologic, renal, and hepatic function.

Exclusion Criteria:

* Subject is diagnosed with brain metastases greater than 28 days prior to Day 1
* Subject received any prior form of cranial radiation and/or neurosurgery for their brain metastases
* Subject's last dose of anti-cancer therapy or investigational therapy was less than or equal to 7 days prior to Day 1
* Subject has a Karnofsky Performance Score of less than 70
* Subject has significant dyspnea requiring supplemental oxygen therapy
* Subject has liver metastases (restaging is not required for known liver metastases)
* Subject has more than 2 sites (organ systems) of metastases from non-small cell lung cancer with the exception of intra-cranial sites of metastases from non-small cell lung cancer, thoracic sites of metastases from non-small cell lung cancer and bone metastases
* Subject has leptomeningeal metastases or subarachnoid spread of tumor
* Subject has unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or prior anti-cancer treatment
* Subject has a known seizure disorder that is uncontrolled, or has seizures occurring greater than or equal to 3 times a week over the past month. Subjects presenting with symptoms of seizures from the brain metastases are eligible; however he/she should receive adequate anti-seizure medication prior to study treatment
* Subject is pregnant or lactating
* Subject has previously been treated with a poly-(ADP-ribose)-polymerase inhibitor as an investigational agent
* Subject has clinically significant and uncontrolled major medical condition(s)
* Subject has a history of another active cancer within the past 5 years except: cervical cancer in situ, in situ carcinoma of the bladder, basal or squamous cell carcinoma of the skin or other cancer in situ that is considered cured

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2012-10-19; Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Giranda, MD, Study Director — AbbVie

REFERENCES:
- [Result] Chabot P, Hsia TC, Ryu JS, Gorbunova V, Belda-Iniesta C, Ball D, Kio E, Mehta M, Papp K, Qin Q, Qian J, Holen KD, Giranda V, Suh JH. Veliparib in combination with whole-brain radiation therapy for patients with brain metastases from non-small cell lung cancer: results of a randomized, global, placebo-controlled study. J Neurooncol. 2017 Jan;131(1):105-115. doi: 10.1007/s11060-016-2275-x. Epub 2016 Sep 21. PMID 27655223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 87 sites in Argentina, Australia, Belgium, Canada, Chile, Czech Republic, Egypt, Finland, France, Hungary, Korea, Norway, Russia, Spain, Taiwan, Ukraine, and the United States.
Pre-assignment Details: Subjects were randomized in a 1:1:1 ratio to one of three treatment groups. Randomization was stratified by graded prognostic assessment (GPA) score (≤ 2.5 versus > 2.5) and neurological symptoms (symptomatic versus asymptomatic).
Period: Overall Study
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT
Started | 102 | 103 | 102
Received Treatment | 101 | 103 | 102
Completed | 0 | 0 | 0
Not Completed | 102 | 103 | 102
Not completed — Adverse Event Related to progression | 6 | 8 | 12
Not completed — Adverse Event Not Related to Progression | 5 | 4 | 4
Not completed — Withdrawal by Subject | 13 | 10 | 10
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Disease Progression | 2 | 4 | 4
Not completed — Progressive Disease Clinical | 7 | 4 | 7
Not completed — Radiographic & Clinical Progression | 16 | 11 | 15
Not completed — Other | 52 | 62 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT | Total
Number analyzed (Participants) | 102 | 103 | 102 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.71) | 59.8 (8.74) | 61.8 (9.08) | 60.6 (9.20)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 68 | 73 | 64 | 205
  ≥ 65 years | 34 | 30 | 38 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 36 | 124
  Male | 56 | 61 | 66 | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 79 | 85 | 66 | 230
  Black | 0 | 2 | 6 | 8
  Asian | 22 | 16 | 28 | 66
  Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 1
  Multirace | 0 | 0 | 2 | 2
Graded Prognostic Assessment (GPA) [Count of Participants; unit: Participants] — A participant's GPA score was the sum total of each of the following prognostic factors, scored as 0, 0.5, or 1:
  * Age, years > 60 years, 50 - 59 years, or < 50 years)
  * Karnofsky Performance Status (< 70, 70 - 80, or 90 - 100)
  * No. of brain metastases (> 3, 2 - 3, or 1)
  * Extracranial metastases (present or absent) The total GPA score could range from 0 to 4 where lower scores indicate a worse prognosis.
  Participants
    ≤ 2.5 | 91 | 91 | 92 | 274
    > 2.5 | 11 | 12 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the number of days from the date of randomization to the date of death. All events of death were included, regardless of whether the event occurred while the participant was still taking study treatment or after treatment was discontinued. If a participant had not died, the data were censored at the date the participant was last known to be alive.
Time Frame: From randomization up to 36 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT
Number analyzed (Participants) | 102 | 103 | 102
days | 185 [137 to 251] | 209 [169 to 264] | 209 [138 to 255]
Statistical Analysis 1: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; The primary analysis used a Hochberg testing procedure to preserve the familywise error rate for multiple comparisons, where the larger P-value for the comparisons of veliparib 50 mg BID + WBRT with placebo BID + WBRT and veliparib 200 mg BID + WBRT with placebo BID + WBRT were compared to an α = 0.05. If statistically significant (P ≤ 0.05), both comparisons were considered significant. If the larger P-value was not statistically significant, the smaller P-value was compared to an α = 0.025; Test type: Superiority; p = 0.933, Log Rank; Log-rank test stratified by graded prognostic assessment (GPA) score (≤ 2.5 or > 2.5) at screening. Nominal P-values were reported
Statistical Analysis 2: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.909, Log Rank; Log-rank test stratified by GPA score (≤ 2.5 or > 2.5) at screening. Nominal P-values were reported
Statistical Analysis 3: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; Test type: Superiority; p = 0.927, Cox proportional hazard model; Cox proportional hazard model stratified by GPA score (≤ 2.5 or > 2.5) at screening. Nominal P-values were reported; Hazard Ratio (HR) = 0.985, 95% CI 2-sided [0.716 to 1.355]
Statistical Analysis 4: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; Test type: Superiority; p = 0.906, Cox proportional hazard model; Cox proportional hazard model stratified by GPA score (≤ 2.5 or > 2.5) at screening. Nominal P-values were reported; Hazard Ratio (HR) = 0.981, 95% CI 2-sided [0.710 to 1.354]

2. Secondary Outcome: Best Tumor Response Rate
Description: Best tumor response rate was calculated as the percentage of participants with a complete response or partial response, as determined by brain scan imaging (magnetic resonance image or computed tomography) by a central imaging vendor. Response was assessed according to the modified bidimensional criteria:
  Complete response required all of the following: complete disappearance of all target and non-target lesions sustained for at least 4 weeks; no new lesions, including no new leptomeningeal disease; no systemic corticosteroid dose.
  Partial response required all of the following: ≥ 50% decrease compared with baseline in the size of all target lesions sustained for at least 4 weeks; no new lesions, including no new leptomeningeal disease and no unequivocal progression of non-target lesions, which, even in presence of stable disease or progressive disease in target lesions, was significant enough to qualify as progression; stable or reduced daily total systemic corticosteroid dose.
Time Frame: From randomization up to 24 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT
Number analyzed (Participants) | 102 | 103 | 102
percentage of participants | 41.2 [31.5 to 51.4] | 36.9 [27.6 to 47.0] | 42.2 [32.4 to 52.3]
Statistical Analysis 1: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; Test type: Superiority; p = 0.535, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by GPA score (≤ 2.5 or > 2.5) at screening
Statistical Analysis 2: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; Test type: Superiority; p = 0.898, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by GPA score (≤ 2.5 or > 2.5) at screening

3. Secondary Outcome: Time to Intracranial Progression (Radiographic)
Description: Time to intracranial progression (radiographic) was defined as the number of days from the date of randomization to the date of the first intracranial progression, as determined by brain scan imaging (magnetic resonance image [MRI]/ computed tomography [CT] scan) by a central imaging vendor. All confirmed events of intracranial progression were included, regardless of whether the event occurred while the participant was still taking study treatment or had previously discontinued study treatment. If the participant did not have a confirmed event of intracranial progression, their data were censored at the date of the last available intracranial progression assessment. Time to intracranial progression (radiographic) was estimated for each treatment group using Kaplan-Meier methodology.
Time Frame: From randomization up to 24 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT
Number analyzed (Participants) | 102 | 103 | 102
days | 259 [184 to NA] — Could not be estimated due to the low number of events. | 226 [147 to 360] | 224 [137 to 358]
Statistical Analysis 1: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; Test type: Superiority; p = 0.314, Log Rank; Log-rank test stratified by GPA score (≤ 2.5 or > 2.5) at screening
Statistical Analysis 2: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; Test type: Superiority; p = 0.536, Log Rank; Log-rank test stratified by GPA score (≤ 2.5 or > 2.5) at screening
Statistical Analysis 3: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; Test type: Superiority; p = 0.313, Cox proportional hazard model; Cox proportional hazard model stratified by GPA score (≤ 2.5 or > 2.5) at screening; Hazard Ratio (HR) = 1.301, 95% CI 2-sided [0.780 to 2.168]
Statistical Analysis 4: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; Test type: Superiority; p = 0.534, Cox proportional hazard model; Cox proportional hazard model stratified by GPA score (≤ 2.5 or > 2.5) at screening; Hazard Ratio (HR) = 1.181, 95% CI 2-sided [0.698 to 1.999]

4. Secondary Outcome: Time to Clinical Brain Metastasis Progression
Description: Time to clinical brain metastases progression was defined as the number of days from randomization to the date of the first experience of clinical brain metastases progression, as assessed by a team of neuro-oncology experts (Event Review Board). All events of clinical brain metastasis progression were included, regardless of whether the event occurred while the participant was still receiving study treatment or had previously discontinued study treatment. If a participant did not have an event of clinical brain metastases progression, their data were censored at the date of the last available clinical disease progression assessment. Time to clinical brain metastasis progression was estimated for each treatment group using Kaplan-Meier methodology.
Time Frame: From randomization up to 24 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT
Number analyzed (Participants) | 102 | 103 | 102
days | 348 [216 to NA] — Could not be estimated due to the low number of events | 286 [192 to NA] — Could not be estimated due to the low number of events | 255 [204 to 342]
Statistical Analysis 1: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; Test type: Superiority; p = 0.864, Log Rank; Log-rank test stratified by GPA score (≤ 2.5 or > 2.5) at screening
Statistical Analysis 2: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; Test type: Superiority; p = 0.301, Log Rank; Log-rank test stratified by GPA score (≤ 2.5 or > 2.5) at screening
Statistical Analysis 3: Comparison: Placebo BID + WBRT vs Veliparib 50 mg BID + WBRT; Test type: Superiority; p = 0.860, Cox proportional hazard model; Cox proportional hazard model stratified by GPA score (≤ 2.5 or > 2.5) at screening; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.626 to 1.754]
Statistical Analysis 4: Comparison: Placebo BID + WBRT vs Veliparib 200 mg BID + WBRT; Test type: Superiority; p = 0.289, Cox proportional hazard model; Cox proportional hazard model stratified by GPA score (≤ 2.5 or > 2.5) at screening; Hazard Ratio (HR) = 1.295, 95% CI 2-sided [0.803 to 2.086]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days following last dose of study drug; median duration of treatment was 15 days.
Arm/Group | Placebo BID + WBRT | Veliparib 50 mg BID + WBRT | Veliparib 200 mg BID + WBRT
Serious Adverse Events (participants affected / at risk) | 39/101 | 31/103 | 36/102
Other Adverse Events (participants affected / at risk) | 78/101 | 76/103 | 77/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID + WBRT (N=101) | Veliparib 50 mg BID + WBRT (N=103) | Veliparib 200 mg BID + WBRT (N=102)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 2
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0
PROCTALGIA (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 2
FATIGUE (General disorders) | 2 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 0 | 1 | 0
PAIN (General disorders) | 3 | 0 | 0
BACTERIAL INFECTION (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
LUNG INFECTION (Infections and infestations) | 2 | 1 | 0
NOSOCOMIAL INFECTION (Infections and infestations) | 1 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0
ORAL FUNGAL INFECTION (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 8 | 3 | 3
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10 | 16
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 1
BRAIN OEDEMA (Nervous system disorders) | 4 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0
DEMENTIA (Nervous system disorders) | 0 | 1 | 0
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 | 0 | 1
HEMIPLEGIA (Nervous system disorders) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0
NERVE COMPRESSION (Nervous system disorders) | 0 | 1 | 0
SEIZURE (Nervous system disorders) | 3 | 0 | 2
STATUS EPILEPTICUS (Nervous system disorders) | 1 | 0 | 0
VASOGENIC CEREBRAL OEDEMA (Nervous system disorders) | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID + WBRT (N=101) | Veliparib 50 mg BID + WBRT (N=103) | Veliparib 200 mg BID + WBRT (N=102)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 4 | 6
CONSTIPATION (Gastrointestinal disorders) | 11 | 10 | 11
DIARRHOEA (Gastrointestinal disorders) | 8 | 8 | 7
NAUSEA (Gastrointestinal disorders) | 29 | 23 | 32
VOMITING (Gastrointestinal disorders) | 14 | 5 | 9
ASTHENIA (General disorders) | 11 | 9 | 13
FATIGUE (General disorders) | 20 | 27 | 21
PYREXIA (General disorders) | 7 | 7 | 4
ORAL CANDIDIASIS (Infections and infestations) | 7 | 3 | 5
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 5 | 5 | 6
DECREASED APPETITE (Metabolism and nutrition disorders) | 14 | 11 | 15
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 | 7 | 4
DIZZINESS (Nervous system disorders) | 11 | 8 | 10
DYSGEUSIA (Nervous system disorders) | 7 | 4 | 2
HEADACHE (Nervous system disorders) | 15 | 18 | 21
ANXIETY (Psychiatric disorders) | 8 | 6 | 2
INSOMNIA (Psychiatric disorders) | 11 | 10 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 10
ALOPECIA (Skin and subcutaneous tissue disorders) | 19 | 15 | 15
RASH (Skin and subcutaneous tissue disorders) | 2 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.